CLINICAL TRIAL: NCT02788578
Title: Peptide Receptor Radionuclide Therapy (PRRT) in Combination With Lanreotide Autogel: A Retrospective Study in Progressive Digestive and Bronchopulmonary Neuroendocrine Neuroendocrine Tumours
Brief Title: A Retrospective Data Analysis of Therapy With PRRT Combined With Lanreotide Autogel® for Neuroendocrine Tumours
Acronym: PRELUDE
Status: Terminated | Type: Observational
Why Stopped: The study terminated prematurely due to insufficient recruitment.
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: F-FR-52030-344
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Neuroendocrine Tumours
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of the PRELUDE study is to describe the use of lanreotide Autogel® (LAN ATG) combined with Peptide Receptor Radionuclide Therapy (PRRT) in the treatment of progressive neuroendocrine tumours located in the lung or in the digestive system as there is currently limited data on these treatments used together for these types of neuroendocrine tumours.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed metastatic well differentiated Neuroendocrine Tumour (NET) (Grade G1 or G2 according to the World Health Organisation 2010 classification): Gastro-entero-pancreatic (GEP) or Bronchopulmonary (BP) primary tumour, or tumour of unknown origin believed to be of GEP origin, if a primary tumour elsewhere was excluded by multiphasic computerised tomography (CT) or magnetic resonance imaging (MRI)
* Disease progression radiologically documented with evaluable imaging (CT or MRI, digital or print-out), performed within 12 months and within 6 months prior to the first PRRT/LAN ATG cycle
* Metastatic- or locally-advanced, hormonal functioning or nonfunctioning GEP-NET or BP-NET;
* Confirmed presence of Somatostatin Receptors (SSTRs) on all target lesions based on positive SSTR scintigraphy (Octreoscan®/99mTC-tektrotyd) or 68Ga SSTR Positron Emission Tomography-Computerised Tomography (PET/CT) imaging, i.e. Grade ≥2 respectively per the Krenning scale or per the modified Krenning scale

Exclusion Criteria:

* Absence of information regarding LAN ATG treatment: dose received, start date, frequency of injections
* No CT or MRI within 12 months and within 6 months preceding the baseline, or at the end of the last PRRT/LAN ATG cycle
* Absence of information on cumulative activity of PRRT with 177 Lutetium (177Lu) DOTATOC or 177Lu-DOTATATE received (at least 500 mCi (equivalent to 18.5 GBq), for the entire therapy)
* PRRT prior to the first combination cycle of PRRT/LAN ATG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) rate according to the central reading using RECIST (Version 1.1) | Approximately 3 to 6 months after the last PRRT/LAN ATG cycle

SECONDARY OUTCOMES:
PFS rate as per RECIST (Version 1.1) | Up to 12 months post-treatment
Best Overall Response as per RECIST (Version 1.1) | Baseline, until disease progression or end of treatment period (generally 3 to 6 months after the last PRRT/LAN ATG cycle) whichever is earlier
Objective Response Rate as per RECIST (Version 1.1) | Approximately 3 to 6 months after the last PRRT/LAN ATG cycle and up to 12 months post-treatment
Change from baseline (i.e. from Day 1 of the first PRRT/LAN ATG cycle prior to any administration) in the presence and in the severity of diarrhoea and flushing, if any | Baseline, approximately 3 to 6 months after the last PRRT/LAN ATG cycle and up to 12 months post-treatment
Change from baseline (i.e. from Day 1 of the first PRRT/LAN ATG cycle prior to any administration) in the tumour biomarker CgA | Baseline, approximately 3 to 6 months after the last PRRT/LAN ATG cycle
Change from baseline (ie from Day 1 of the first PRRT/LAN ATG cycle prior to any administration) in body weight | Baseline, approximately 3 to 6 months after the last PRRT/LAN ATG cycle and up to 12 months post-treatment
Incidence of nephrotoxicity, haematotoxicity and hepatotoxicity events (based on a predefined list of disorders) | Baseline, approximately 3 to 6 months after the last PRRT/LAN ATG cycle and up to 12 months post-treatment
Incidence of vomiting (during infusion only) | Approximately 3 to 6 months after the last PRRT/LAN ATG cycle

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (12):
- Peter MacCallum Cancer Centre, East Melbourne, Australia
- France (2):
  - IUCT Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - Zentralklinil Bad Berka, Bad Berka
  - Charité, Berlin
  - Klinikum rechts der Usar, München
- Italy (2):
  - Unversità degli Studi di Messina, Messina
  - IEO Institutio Europeo di Oncologia, Milan
- United Kingdom (4):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Kings College Hospital, London
  - Royal Free Hospital London, London
  - The Christie NHS Foundation Trust, Manchester

REFERENCES:
- [Derived] Prasad V, Srirajaskanthan R, Toumpanakis C, Grana CM, Baldari S, Shah T, Lamarca A, Courbon F, Scheidhauer K, Baudin E, Truong Thanh XM, Houchard A, Dromain C, Bodei L. Lessons from a multicentre retrospective study of peptide receptor radionuclide therapy combined with lanreotide for neuroendocrine tumours: a need for standardised practice. Eur J Nucl Med Mol Imaging. 2020 Sep;47(10):2358-2371. doi: 10.1007/s00259-020-04712-2. Epub 2020 Feb 15. PMID 32062681